CLINICAL TRIAL: NCT05332171
Title: Examination Of Exercise Adherence İn Lung Cancer Patients Given Calisthenic Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Kardelen HATIMOĞULLARI, physiotherapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/026
Record Dates: First submitted 2022-04-05; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Exercise Addiction; Lung Cancer
Keywords: Lung Cancer; Pulmonary Rehabilitation; calisthenic exercise; exercise adherence
MeSH Terms: conditions — Lung Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: It is aimed to evaluate patients with Lung Cancer who meet the inclusion criteria of the study. Individuals will be randomly assigned to physical activity counseling and training groups. The number of participants in the groups will be determined by power analysis.
  Criteria for inclusion in the study;
  * Patients whose chemotherapy and radiotherapy has ended, at least 6 months and maximum 5 years after surgery
  * Being between the ages of 18-65
  * 3 and 5 years according to the Modified Borg Scale Patients with severe fatigue Exclusion criteria;
  * Uncontrollable hypertension, diabetes mellitus, heart failure and atrial fibrillation
  * Any acute infection during the evaluation
  * Orthopedic, neurological, psychological, etc., which will limit the evaluations. with problems
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical activity counseling (No Intervention): Home exercises will be taught to the physical activity counseling group and will be followed up under the supervision of a physiotherapist with weekly controls. Evaluation will be done before and after treatment.
- training group (Active Comparator): Breathing exercises and calisthenic exercises will be taught to the training group, and they will be followed under the supervision of a physiotherapist for 8 weeks, 3 days a week. Evaluations will be made before and after treatment. Individuals in the calisthenic exercise group will be given exercise training at the level of 65%-80% of the maximal heart rate for 30-40 minutes, 3 days a week for 8 weeks.
  Interventions: Behavioral: Pyhsiohterapy and rehabilitation

INTERVENTIONS:
Behavioral: Pyhsiohterapy and rehabilitation — Before starting the exercise program, 10 repetitive warm-up exercises will be given including the lower and upper extremities and distal joints. The exercises will be started with 5 repetitions in the first week. Depending on the patient's tolerance, the intensity of the exercise will be increased as 10 repetitions, 15 repetitions and 20 repetitions, and optional rest will be allowed between exercises. It is aimed that the patients reach 20 repetitions in the 6th week at the latest.
  Arms: training group

SUMMARY:
Cancer treatments usually include surgery, chemotherapy, radiation therapy, hormone therapy, and/or a combination of these methods. These treatments cause many physical and psychological effects that interfere with functional independence, performing activities of daily living, and healthy quality of life. Mostly, depending on cancer and its treatment; Cognitive function, sleep pattern, functional capacity, pain state and bone mineral density are affected. Exercise compliance is the degree to which an individual's behavior is consistent with the health care provider's advice and treatment plan. According to the World Health Organization, compliance is "a measure of a person's behavior (such as following a recommended exercise program, monitoring drug intake, etc.). ) as a response to complying with recommendations deemed appropriate by health care professionals''. In the field of rehabilitation too, compliance is increasingly used in relation to the self-management of patients' health. It has been stated in the studies that the level of compliance with the recommended home exercise is generally low, which limits the benefits of exercise programs.

DETAILED DESCRIPTION:
This study is a cross-sectional study. Lung cancer patients who applied to the Oncology Service and met the inclusion criteria will be included in the study. Patients will be randomly assigned to physical activity counseling and education groups.

Within the scope of the study, exercise compliance will be examined in patients with lung cancer who are given calisthenic exercise.

Participants will be evaluated before treatment, their functional capacities will be determined, their compliance with exercise, fatigue levels, pain levels, cognitive status, sleep and quality of life will be evaluated with questionnaires.

Home exercises will be taught to the physical activity counseling group and will be followed up under the supervision of a physiotherapist with weekly controls. Breathing exercises and calisthenic exercises will be taught to the training group, and participants will be followed under the supervision of a physiotherapist for 8 weeks, 3 days a week. Evaluations will be made before and after the treatment.

Individuals who do not agree to / give up participating in the study will be able to leave the study voluntarily.

All information belonging to individuals will be protected according to the personal data protection law.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose chemotherapy and radiotherapy has ended, at least 6 months and maximum 5 years after surgery
* Being between the ages of 18-65
* 3 and 5 years according to the Modified Borg Scale Patients with severe fatigue

Exclusion Criteria:

* Uncontrollable hypertension, diabetes mellitus, heart failure and atrial fibrillation
* Any acute infection during the evaluation
* Orthopedic, neurological, psychological, etc., which will limit the evaluations. with problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Exercise compliance of patients with lung cancer who are given calisthenic exercise increases | 8 week
  Exercise compliance increases in patients who are given calisthenic exercises accompanied by a physiotherapist.

SECONDARY OUTCOMES:
The functional capacity of patients with lung cancer who are given calisthenic exercise increases. | 8 week
  The functional capacity of patients with lung cancer who are given calisthenic exercises under the guidance of a physiotherapist increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Univercity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided